CLINICAL TRIAL: NCT04257201
Title: Mushroom Ingestion Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Mushroom Council (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Principal Investigator, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB-2019-645
Record Dates: First submitted 2019-12-18; First posted 2020-02-05 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Diet, Healthy
Keywords: Mediterranean; Mushrooms; Metabolomics

STUDY DESIGN:
Intervention Model Description: For this randomized crossover study, subjects will consume 5 test meals varying in mushroom content, each separated by a minimum of 10 days (Figure 1). For 3 days prior to each testing day participants will be provided with and instructed to exclusively consume a low-antioxidant "run-in" diet (low fruit, vegetable, and spice diet) to minimize background concentrations of potential test food-derived compounds of interest. On test days, participants will consume a standardized mixed-macronutrient meal (500 kcal, 75g CHO, 15g Protein, 15g Fat) containing 1) no mushrooms (control), 2) 84 g of raw white button mushrooms served cooked; 3) 168 g of raw white button mushrooms served cooked; 4) 84 g of raw yellow oyster mushrooms served cooked; or 5) 168 g of raw yellow oyster mushrooms served cooked. Between each run-in diet/testing period, participants will consume their usual, unrestricted self-selected diets for a minimum of 7 days.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control -- no mushrooms (Active Comparator): Subjects will be randomized to consume a test day salad with 0 g, 84 g (yellow oyster or white button) or 168 g (yellow or white button) mushrooms. Mushrooms will be cooked prior to serving.
  Interventions: Other: Control
- Yellow Oyster -- 84 g (Experimental): Subjects will be randomized to consume a test day salad with 0 g, 84 g (yellow oyster or white button) or 168 g (yellow or white button) mushrooms. Mushrooms will be cooked prior to serving.
  Interventions: Other: Yellow Oyster -- 84 g
- Yellow Oyster -- 168 g (Experimental): Subjects will be randomized to consume a test day salad with 0 g, 84 g (yellow oyster or white button) or 168 g (yellow or white button) mushrooms. Mushrooms will be cooked prior to serving.
  Interventions: Other: Yellow Oyster -- 168 g
- White button -- 84 g (Experimental): Subjects will be randomized to consume a test day salad with 0 g, 84 g (yellow oyster or white button) or 168 g (yellow or white button) mushrooms. Mushrooms will be cooked prior to serving.
  Interventions: Other: White button -- 84 g
- White button 168 g (Experimental): Subjects will be randomized to consume a test day salad with 0 g, 84 g (yellow oyster or white button) or 168 g (yellow or white button) mushrooms. Mushrooms will be cooked prior to serving.
  Interventions: Other: White button -- 168 g

INTERVENTIONS:
Other: Yellow Oyster -- 84 g — Participants will consume the standardized test day salad plus 84 g (raw weight) mushrooms. Mushrooms will be cooked prior to being served
  Arms: Yellow Oyster -- 84 g
Other: Yellow Oyster -- 168 g — Participants will consume the standardized test day salad plus 168 g (raw weight) mushrooms. Mushrooms will be cooked prior to being served
  Arms: Yellow Oyster -- 168 g
Other: White button -- 84 g — Participants will consume the standardized test day salad plus 84 g (raw weight) mushrooms. Mushrooms will be cooked prior to being served
  Arms: White button -- 84 g
Other: White button -- 168 g — Participants will consume the standardized test day salad plus 168 g (raw weight) mushrooms. Mushrooms will be cooked prior to being served
  Arms: White button 168 g
Other: Control — Participants will consume the standardized test day salad only
  Arms: Control -- no mushrooms

SUMMARY:
The investigators propose to determine the effect of consuming 0, 1 or 2 servings of white button (Agaricus bisporus; most popular, lower ergothioneine) or yellow oyster (Pleurotus citrinopileatus; higher ergothioneine) mushrooms on postprandial changes in plasma levels and urinary excretions of mushroom-specific compounds.

DETAILED DESCRIPTION:
The investigators hypothesize that consuming different mushroom varieties will elicit distinct postprandial nutrimetabolomic profiles in the plasma and urine and that the amount of metabolites present will increase with the servings of mushrooms. Measuring ergothioneine in the plasma will provide a quantitative outcome to document the postprandial responses to consuming the test meals. The nutrimetabolomic related outcomes are exploratory and have not been documented in human research.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* age 30-69 y;
* BMI: 25.0-34.9 kg/m2;
* Not severely or extremely depressed (Beck's Depression Inventory score ≤30)
* Total cholesterol <240 mg/dL, low-density lipoprotein cholesterol <160 mg/dL, triglycerides <400 mg/dL, fasting glucose <110 mg/dL;
* Systolic/diastolic blood pressure <140/90 mm Hg;
* Body weight stable for 3 months prior (± 3 kg);
* Stable physical activity regimen 3 months prior;
* Medication use stable for 6 months prior;
* Non-smoking;
* Non-diabetic;
* Not acutely ill;
* Females not pregnant or lactating;
* Participants must be willing and able to consume the prescribed diets and travel to testing facilities.

Exclusion Criteria:

* BMI <25 or >35;
* Severely depressed (Beck's Depression Inventory score >30);
* Total cholesterol >240 mg/dL, low-density lipoprotein cholesterol >160 mg/dL, triglycerides >400 mg/dL, fasting glucose >110 mg/dL;
* Body weight changes in previous 3 months (±3 kg);
* Changes in physical activity regimen in the previous 3 months;
* Medication changes in the previous 6 months;
* Smoking;
* Diabetic;
* Acute illness;
* Pregnant or lactating;
* Allergic to mushrooms

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Change in plasma glucose | 5 hours
  Plasma will be assessed for glucose values prior to salad consumption and in response to the test day meal
Change in plasma insulin | 5 hours
  Plasma will be assessed for insulin values prior to salad consumption and in response to the test day meal
Plasma metabolomics | 5 hours
  Plasma will be assessed for metabolomics (i.e. ergothioneine) via reverse phase liquid chromatography/mass spectrometry
Plasma ergothioneine | 5 hours
  Plasma will be assessed for ergothioneine concentration, a compound unique to mushrooms
Plasma triglycerides | 5 hours
  Plasma will be assessed for triglyceride values at the time of salad consumption and at each hour for 5 hours after salad consumption

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Campbell, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States